CLINICAL TRIAL: NCT03312751
Title: An Open-label, Single Arm, Multicenter Study to Broaden Access to Emapalumab, an Anti-Interferon Gamma (Anti-IFNγ) Monoclonal Antibody, and to Assess Its Efficacy, Safety, Impact on Quality of Life, and Long-term Outcome in Pediatric Patients With Primary Hemophagocytic Lymphohistiocytosis
Brief Title: Study to Assess the Efficacy and Safety of Emapalumab in Primary Haemophagocytic Lymphohistiocytosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-0501-09
Record Dates: First submitted 2017-10-05; First posted 2017-10-18 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Primary Hemophagocytic Lymphohistiocytosis
Keywords: Interferon-gamma; NI-0501; primary HLH; emapalumab
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Emapalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emapalumab (Experimental)
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Emapalumab will be administered by intravenous infusion, twice weekly.

SUMMARY:
The purpose of this study is to expand the knowledge on the efficacy and safety of emapalumab (previously known as NI-0501) as a treatment for primary haemophagocytic lymphohistiocytosis (HLH) patients, including on long-term outcomes and quality of life assessments. Emapalumab can be administered as the first-line therapy to patients not previously treated with the current standard of care, or can be given to patients who have either failed or were unable to tolerate the available standard of care.

Emapalumab is to be administered until the start of conditioning for hematopoietic stem cell transplantation (HSCT), with an anticipated duration ranging from a minimum of 4 weeks to approximately 12 weeks and not exceeding 6 months.

After treatment completion, patients will continue in the study for long-term follow-up until 1 year after either HSCT or last emapalumab infusion (if HSCT is not performed).

ELIGIBILITY:
Main Inclusion Criteria:

* Primary HLH patients with active disease.
* Treatment naïve patients or patients having already received HLH conventional therapy, but having not responded, not achieved a satisfactory response or worsened, or reactivated, or are unable to tolerate current standard of care.
* Informed consent signed by the patient or by the patient's legally authorized representative.
* Received guidance on contraception.

Main Exclusion Criteria:

* Diagnosis of secondary HLH consequent to a proven rheumatic, metabolic or neoplastic disease.
* Active mycobacteria, Histoplasma capsulatum, Shigella, Salmonella, Campylobacter or Leishmania infections.
* Evidence of latent tuberculosis.
* Presence of malignancy.
* Concomitant disease or malformation severely affecting cardiovascular, pulmonary, central nervous system (CNS), liver, or renal function, that in the opinion of the Investigator may significantly affect the likelihood to respond to treatment and/or the assessment of emapalumab safety and/or efficacy.
* History of hypersensitivity or allergy to any component of the study regimen.
* Receipt of a BCG vaccine within 12 weeks prior to Screening.
* Receipt of a live or attenuated-live (other than BCG) vaccine within 6 weeks prior to Screening.
* Pregnant or lactating female patients.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (10):
  - Phoenix Children Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. duPont Hospital for Children - Nemours Center for Cancer and Blood Disorders - Division of Pediatric Hematology Oncology, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Spectrum Health Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Texas Children's Hospital - Feigin Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Hopital Ste-Justine Research Center, Montreal
  - Hospital for Sick Children, Toronto
  - Children's and Women's Health Centre of British Columbia, Vancouver
- Germany (3):
  - Universitätsklinikum Essen, Essen
  - Medical Center- University of Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Eppendorf, Hamburg
- Italy (4):
  - Istituto Giannina Gaslini, Genova
  - Fondazione MBBM, Ospedale San Gerardo, Monza
  - Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale della Donna e del Bambino, Verona
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Niño Jesús, Madrid
- Karolinska University Hospital Huddinge, Stockholm, Sweden
- University Children's Hospital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Leeds Children's Hospital, Leeds
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- All-treated Analysis Set - Treatment naïve: The All-treated analysis set included all patients who received any part of an infusion of study drug. The All-treated analysis set was the primary analysis set for efficacy endpoints and was used for safety and PK/PD endpoints. Details are reported in this arm for patients in the All-treated analysis set who were naïve to HLH treatment.
- All-treated Analysis Set - Treatment Experienced: The All-treated analysis set included all patients who received any part of an infusion of study drug. The All-treated analysis set was the primary analysis set for efficacy endpoints and was used for safety and PK/PD endpoints. Details are reported in this arm for patients in the All-treated analysis set who have received conventional HLH therapy (as per site standard of care), without having obtained a satisfactory response according to the Investigator or having shown signs of intolerance to previous HLH therapy.
Period: Overall Study
Arm/Group | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Started | 16 | 19
Completed | 9 | 9
Not Completed | 7 | 10
Not completed — Death | 7 | 9
Not completed — Study discontinuation due to other reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 19 | 35
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 12 | 18 | 30
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 6 | 12 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Body Weight (kg) [Mean (Standard Deviation); unit: kg] — Baseline observation is the last observation recorded prior to the first dose of emapalumab.
  kg | 9.599 (10.5915) | 13.946 (14.4351) | 11.959 (12.8309)
Height/Length (cm) [Mean (Standard Deviation); unit: cm] — Baseline observation is the last observation recorded prior to the first dose of emapalumab.
  cm | 67.02 (27.416) | 83.41 (37.790) | 75.96 (34.003)
Body Surface Area (m^2) [Mean (Standard Deviation); unit: m^2] — Baseline observation is the last observation recorded prior to the first dose of emapalumab.
  m^2 | 0.415 (0.3022) | 0.564 (0.4141) | 0.497 (0.3698)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response at Week 8 or End of Treatment (if Earlier)
Description: The overall response rate (ORR) of patients achieving either Complete or Partial Response or HLH Improvement, at Week 8 or EOT (whichever occurs earlier).
Time Frame: Up to Week 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All-treated Analysis Set: The All-treated analysis set included all patients who received any part of an infusion of study drug. The All-treated analysis set was the primary analysis set for efficacy endpoints and was used for safety and PK/PD endpoints.
- All-treated Analysis Set - Treatment naïve: Patients in the All-treated analysis set who were naïve to HLH treatment.
- All-treated Analysis Set - Treatment Experienced: Patients in the All-treated analysis set who have received conventional HLH therapy (as per site standard of care), without having obtained a satisfactory response according to the Investigator or having shown signs of intolerance to previous HLH therapy.
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Percentage of participants | 62.9 [44.9 to 78.5] | 50.0 [24.7 to 75.3] | 73.7 [48.8 to 90.9]
Statistical Analysis 1: Comparison: All-treated Analysis Set; The primary efficacy endpoint was analyzed with an exact binomial test to evaluate the null hypothesis that the Overall Response Rate was, at most, 40%. This test was performed at the one sided 0.025 significance level; Test type: Superiority; p = 0.0053, Exact binomial; Overall response rate = 62.9, 95% CI 2-sided [44.9 to 78.5]
Statistical Analysis 2: Comparison: All-treated Analysis Set - Treatment naïve; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2839, Exact binomial
Statistical Analysis 3: Comparison: All-treated Analysis Set - Treatment Experienced; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0031, Exact binomial

2. Secondary Outcome: Overall Survival at End of Study
Description: Number of patients surviving to the end of the study.
Time Frame: Up to 18 months
Population: 'All-treated analysis set - treatment experienced' includes a censored observation for 1 patient who discontinued the study early.
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants
  Alive at end of study | 19 | 9 | 10
  Early discontinuation | 1 | 0 | 1

3. Secondary Outcome: Overall Survival to HSCT
Description: Number of patients surviving to HSCT.
Time Frame: From start of treatment to HSCT or from start of treatment until 1 year after EOT for patient who did not undergo HSCT
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants | 25 | 12 | 13

4. Secondary Outcome: Overall Survival for Patients Receiving HSCT
Description: Number of patients surviving post HSCT.
Time Frame: Up to 1 year post HSCT
Population: All-treated analysis includes total number or patients who received HSCT.
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 23 | 11 | 12
Participants | 17 | 8 | 9

5. Secondary Outcome: Event-free Survival
Description: Number of patients experiencing event-free survival, the duration of which was defined as time from HSCT to date of (whichever occurs first): death from any cause, graft failure, or HLH reactivation.
Time Frame: Up to 1 year post HSCT
Population: Analysis population based on the number of patients with HSCT.
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 23 | 11 | 12
Participants | 16 | 8 | 8

6. Secondary Outcome: Overall Response at Start of Conditioning
Description: Number of patients achieving either a Complete or Partial Response or HLH Improvement, at start of conditioning (or at last emapalumab infusion if HSCT is not performed).
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants
  Complete response | 4 | 3 | 1
  Partial response | 11 | 5 | 6
  HLH improvement | 1 | 0 | 1
  No response | 19 | 8 | 11

7. Secondary Outcome: Duration of Response
Description: Duration of response, i.e., maintenance of the response achieved at any time during the study (with censoring time at start of conditioning for patients with no event) calculated only for patients showing confirmed overall response. Summarized by number of patients experiencing each category of response duration.
Time Frame: Up to 18 months
Population: Only patients showing at least one maintained response were included. Duration of response is defined as maintenance of response for at least 4 days, achieved at any time during the study until EOT. Patients who do not achieve at least HLH improvement between the date of first dose and EOT are excluded from the analysis. For both first response and loss of response, persistence for at least 4 days is required, otherwise the next response/loss of response period will be considered.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 28 | 12 | 16
days | 61 [29.0 to NA] — NA explanation: The upper CI could not be calculated as there were not enough subjects that had a response and subsequently lost that response in the observed time period | 40 [19.0 to NA] — NA explanation: The upper CI could not be calculated as there were not enough subjects that had a response and subsequently lost that response in the observed time period | 61 [21.0 to NA] — NA explanation. The upper CI could not be calculated as there were not enough subjects that had a response and subsequently lost that response in the observed time period

8. Secondary Outcome: Time to Response
Description: Time to first response at any time during the study.
Time Frame: Up to 18 months
Population: Only patients with a response were included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 28 | 12 | 16
days | 4 [4.0 to 13.0] | 5 [4.0 to 21.0] | 4 [4.0 to 30.0]

9. Secondary Outcome: Number of Patients Reducing Glucocorticoids by 50% or More of the Baseline Dose During Emapalumab Treatment
Description: Number of patients able to reduce glucocorticoids by 50% or more of the baseline dose during emapalumab treatment.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants | 15 | 8 | 7

10. Secondary Outcome: Number of Patients Proceeding to HSCT
Description: Number of patients able to proceed to HSCT when deemed indicated.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants | 23 | 11 | 12

11. Secondary Outcome: Quality of Life Assessed Through PedsQL™, Pediatric Quality of Life Inventory™
Description: Assessment of the quality of life using the PedsQL "Pediatric Quality of Life Inventory". The PedsQL uses a 100-point scale ranging from 0 to 100 with higher values indicating better quality of life.
Time Frame: Up to 6 months
Population: Results from the PedsQL were not available for all patients; in addition, due to the age and treatment history of patients, not all age categories were represented in each of the analysis sets.
Measure: Mean (Standard Deviation); unit: scale on a score
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 20 | 6 | 14
scale on a score
  Change from Baseline at EOT/Week 8 - 1-12 months: number analyzed (Participants) | 11 | 5 | 6
  Change from Baseline at EOT/Week 8 - 1-12 months | 0.208 (18.0737) | -6.514 (14.8977) | 5.810 (19.8220)
  Change from Baseline at EOT/Week 8 - 13-24 months: number analyzed (Participants) | 3 | 0 | 3
  Change from Baseline at EOT/Week 8 - 13-24 months | 0.794 (4.8152) |  | 0.794 (4.8152)
  Change from Baseline at EOT/Week 8 - 2-4 years: number analyzed (Participants) | 3 | 0 | 3
  Change from Baseline at EOT/Week 8 - 2-4 years | 8.469 (9.6897) |  | 8.469 (9.6897)
  Change from Baseline at EOT/Week 8 - 5-7 years: number analyzed (Participants) | 0 | 0 | 0
  Change from Baseline at EOT/Week 8 - 8-12 years: number analyzed (Participants) | 1 | 1 | 0
  Change from Baseline at EOT/Week 8 - 8-12 years | 15.978 | 15.978 |
  Change from Baseline at EOT/Week 8 - 13-18 years: number analyzed (Participants) | 2 | 0 | 2
  Change from Baseline at EOT/Week 8 - 13-18 years | -7.862 (13.4760) |  | -7.862 (13.4760)

12. Secondary Outcome: Quality of Life Assessed Through Behavioral, Affective and Somatic Experiences Scales (BASES)
Description: Assessment of the quality of life using the BASES questionnaire, which is a validated 38-item questionnaire; a reduced nonvalidated 22-item version of the questionnaire is used in an exploratory nature for the secondary endpoint.
  Subscale scores were calculated using a 5-point Likert scale from 1 to 5 for all questions. Scores for all questions in each subscale were added up and divided by the number of patients in the analysis population to reach the mean score. Subscale scores were calculated for the following domains:
  * Physical Discomfort (5 questions, '1' = best response, total range 5-25)
  * Cooperation/Compliance (5 questions, '1' = best response, total range 5-25)
  * Mood/Behavior (7 questions, '5' = best response, total range 7-35)
  * Quality of Interactions (3 questions, '1' = best response, total range 3-15)
  * Activity/Sleep (2 questions, '5' = best response for patient's activity level and '1' = best response for patient's sleeping, total range 2-10)
Time Frame: Up to 6 months
Population: Assessment completed at the end of treatment for those who proceeded/were planned to proceed to HSCT.
Measure: Mean (Standard Deviation); unit: scale on a score
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 15 | 7 | 8
scale on a score
  Physical discomfort | 10.0 (3.57) | 9.4 (2.99) | 10.5 (4.14)
  Cooperation/compliance | 9.3 (3.02) | 9.6 (2.76) | 9.1 (3.4)
  Mood/behavior | 20.4 (8.82) | 15.1 (8.88) | 25.0 (6.02)
  Quality of interactions | 5.8 (2.34) | 6.1 (2.48) | 5.5 (2.33)
  Activity | 3.1 (1.22) | 2.7 (0.95) | 3.4 (1.41)
  Sleep: number analyzed (Participants) | 11 | 5 | 6
  Sleep | 2.1 (1.04) | 1.8 (1.10) | 2.3 (1.03)

13. Secondary Outcome: Incidence, Severity, Causality and Outcomes of AEs (Serious and Non-serious)
Description: Incidence of adverse events. SAE = serious adverse event; TEAE = treatment-emergent adverse event
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants
  Non-TEAEs | 15 | 5 | 10
  TEAEs | 35 | 16 | 19
  TEAEs related to study drug | 9 | 3 | 6
  Mild TEAEs | 30 | 12 | 18
  Moderate TEAEs | 27 | 12 | 15
  Severe TEAEs | 31 | 15 | 16
  TEAEs leading to discontinuation of study drug | 7 | 3 | 4
  TEAEs with an outcome of death | 16 | 7 | 9
  Serious TEAEs | 32 | 16 | 16
  Treatment-emergent SAEs related to study drug | 4 | 2 | 2
  TEAEs with infections | 29 | 14 | 15
  Mild infections | 21 | 10 | 11
  Moderate infections | 15 | 8 | 7
  Severe infections | 16 | 7 | 9
  TEAEs with infusion-related reactions | 7 | 3 | 4

14. Secondary Outcome: Evolution of Laboratory Parameters Change From Baseline to EOT/Week 8
Description: Number of patients experiencing shifts from baseline in the following relevant laboratory parameters are reported:
  * Biochemistry: glucose ferritin, C-reactive protein (CRP), liver function (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma glutamyl transferase [γGT], lactate dehydrogenase [LDH], bilirubin, renal function (albumin, creatinine, urea, urea nitrogen), triglycerides
  * Complete blood count: basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes, hematocrit, hemoglobin, large unstained cells, lymphocytes, lymphocytes/leukocytes, monocytes, monocytes/leukocytes, neutrophils band form, neutrophils band form/leukocytes, platelets, erythrocytes, leukocytes
  * Coagulation tests (activated partial thromboplastin time [aPTT], aPTT ratio, prothrombin time, prothrombin international normalized ratio [INR]), D-dimer, fibrinogen
Time Frame: To Week 8 or End of treatment if before Week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants
  Albumin: low to within | 6 | 3 | 3
  Albumin: within to low | 2 | 0 | 2
  Alkaline phosphatase: low to within | 5 | 1 | 4
  Alkaline phosphatase: within to low | 8 | 5 | 3
  Alkaline phosphatase: high to within | 2 | 1 | 1
  Alanine aminotransferase: within to high | 3 | 1 | 2
  Alanine aminotransferase: high to within | 8 | 6 | 2
  Aspartate aminotransferase: within to high | 3 | 0 | 3
  Aspartate aminotransferase: high to low | 1 | 1 | 0
  Aspartate aminotransferase: high to within | 8 | 5 | 3
  Bilirubin: within to low | 1 | 1 | 0
  Bilirubin: within to high | 1 | 0 | 1
  Bilirubin: high to within | 4 | 2 | 2
  Creatinine: low to within | 1 | 0 | 1
  Creatinine: within to low | 5 | 1 | 4
  Creatinine: within to high | 1 | 0 | 1
  Creatinine: high to within | 2 | 1 | 1
  C-reactive protein: within to high | 6 | 2 | 4
  C-reactive protein: high to within | 4 | 1 | 3
  Ferritin: high to low | 1 | 1 | 0
  Ferritin: high to within | 5 | 3 | 2
  γGT: within to high | 3 | 1 | 2
  γGT: high to within | 4 | 3 | 1
  Glucose: within to high | 2 | 2 | 0
  Glucose: high to within | 8 | 4 | 4
  Lactate dehydrogenase: low to within | 1 | 0 | 1
  Lactate dehydrogenase: within to high | 4 | 2 | 2
  Lactate dehydrogenase: high to within | 8 | 5 | 3
  Triglycerides: within to high | 1 | 0 | 1
  Triglycerides: high to within | 5 | 3 | 2
  Urea: within to low | 5 | 2 | 3
  Urea: within to high | 4 | 2 | 2
  Urea: high to within | 4 | 1 | 3
  Urea nitrogen: low to within | 1 | 1 | 0
  Urea nitrogen: within to low | 1 | 1 | 0
  Urea nitrogen: within to high | 1 | 1 | 0
  Basophils: low to within | 1 | 0 | 1
  Basophils: within to high | 1 | 0 | 1
  Basophils: high to within | 1 | 1 | 0
  Basophils/leukocytes: high to within | 1 | 1 | 0
  Eosinophils: low to within | 3 | 1 | 2
  Eosinophils: within to low | 1 | 1 | 0
  Eosinophils/leukocytes: within to high | 2 | 1 | 1
  Hematocrit: low to within | 9 | 4 | 5
  Hematocrit: within to low | 5 | 2 | 3
  Hemoglobin: low to within | 9 | 5 | 4
  Hemoglobin: low to high | 1 | 0 | 1
  Hemoglobin: within to low | 5 | 1 | 4
  Large unstained cells: high to within | 1 | 1 | 0
  Lymphocytes: low to within | 4 | 2 | 2
  Lymphocytes: within to low | 6 | 3 | 3
  Lymphocytes: within to high | 1 | 1 | 0
  Lymphocytes: high to within | 1 | 1 | 0
  Lymphocytes/leukocytes: within to high | 1 | 1 | 0
  Lymphocytes/leukocytes: within to low | 4 | 2 | 2
  Lymphocytes/leukocytes: high to within | 2 | 2 | 0
  Monocytes: low to within | 6 | 2 | 4
  Monocytes: low to high | 3 | 0 | 3
  Monocytes: within to low | 2 | 1 | 1
  Monocytes: within to high | 2 | 2 | 0
  Monocytes: high to within | 2 | 0 | 2
  Monocytes/leukocytes: within to high | 3 | 3 | 0
  Monocytes/leukocytes: high to within | 1 | 1 | 0
  Neutrophils band form: low to within | 9 | 3 | 6
  Neutrophils band form: within to low | 2 | 1 | 1
  Neutrophils band form: within to high | 2 | 0 | 2
  Neutrophils band form: high to within | 1 | 1 | 0
  Neutrophils band form/leukocytes: low to within | 2 | 1 | 1
  Neutrophils band form/leukocytes: within to low | 1 | 1 | 0
  Neutrophils band form/leukocytes: within to high | 1 | 1 | 0
  Platelets: low to within | 5 | 2 | 3
  Platelets: low to high | 2 | 2 | 0
  Platelets: within to low | 3 | 1 | 2
  Platelets: within to high | 1 | 0 | 1
  Platelets: high to within | 1 | 0 | 1
  Erythrocytes: low to within | 8 | 4 | 4
  Erythrocytes: within to low | 4 | 2 | 2
  Erythrocytes: within to high | 1 | 0 | 1
  Leukocytes: low to within | 9 | 2 | 7
  Leukocytes: low to high | 1 | 1 | 0
  Leukocytes: within to low | 4 | 3 | 1
  Leukocytes: high to within | 1 | 1 | 0
  aPTT: low to within | 2 | 1 | 1
  aPTT: within to low | 4 | 2 | 2
  aPTT: within to high | 3 | 1 | 2
  aPTT: high to within | 4 | 3 | 1
  aPTT ratio: low to within | 2 | 0 | 2
  aPTT ratio: within to low | 1 | 0 | 1
  aPTT ratio: within to high | 2 | 0 | 2
  aPTT ratio: high to within | 2 | 2 | 0
  D-dimer: within to high | 4 | 0 | 4
  D-dimer: high to within | 6 | 4 | 2
  Fibrinogen: low to within | 13 | 6 | 7
  Fibrinogen: low to high | 1 | 0 | 1
  Fibrinogen: within to low | 2 | 1 | 1
  Fibrinogen: within to high | 2 | 1 | 1
  Fibrinogen: high to within | 3 | 1 | 2
  Prothrombin time: within to high | 3 | 1 | 2
  Prothrombin time: high to within | 6 | 3 | 3
  Prothrombin INR: within to high | 1 | 0 | 1
  Prothrombin INR: high to low | 1 | 1 | 0
  Prothrombin INR: high to within | 4 | 2 | 2

15. Secondary Outcome: Number of Patients Who Discontinued Emapalumab Treatment
Description: Number of patients who discontinued emapalumab treatment for safety reasons.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants | 7 | 3 | 4

16. Other Pre Specified Outcome: Serum Concentrations of Emapalumab
Description: The serum concentration of emapalumab will be measured as a function of time to determine the emapalumab PK profile.
Time Frame: Up to Week 8, with data presented at Baseline and EOT/W8
Population: The number of participants analyzed at each timepoint reflects the number of participants who provided samples.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
ng/mL
  Emapalumab serum concentration at Baseline pre-dose: number analyzed (Participants) | 34 | 15 | 19
  Emapalumab serum concentration at Baseline pre-dose | 14.311 (50.2717) | 12.899 (49.9589) | 15.425 (51.8562)
  Emapalumab serum concentration at EOT/Week 8 pre-dose: number analyzed (Participants) | 31 | 13 | 18
  Emapalumab serum concentration at EOT/Week 8 pre-dose | 258337.456 (231412.7632) | 295521.381 (296009.6195) | 231482.400 (175589.7297)
  Emapalumab serum concentration at EOT/Week 8 post-dose: number analyzed (Participants) | 2 | 1 | 1
  Emapalumab serum concentration at EOT/Week 8 post-dose | 142338.620 (89464.1682) | 205599.340 (NA) — Not calculable | 79077.900 (NA) — Not calculable

17. Other Pre Specified Outcome: Change in Pharmacodynamic Parameters
Description: Levels (in ng/L) of total IFNγ (interferon gamma), markers of its neutralization (CXCL9 and CXCL10), and sCD25.
Time Frame: Up to 18 months with data presented at Baseline and EOT/W8
Population: The number of participants analyzed at each timepoint reflects the number of participants who provided samples.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
ng/L
  Total IFNγ at baseline: number analyzed (Participants) | 34 | 15 | 19
  Total IFNγ at baseline | 1112.681 (2393.9753) | 1356.191 (2550.8868) | 920.436 (2314.6502)
  Total IFNγ at EOT/Week 8: number analyzed (Participants) | 31 | 13 | 18
  Total IFNγ at EOT/Week 8 | 25708.836 (41775.8890) | 39233.258 (60957.7563) | 15941.198 (14695.7764)
  CXCL10 at baseline: number analyzed (Participants) | 33 | 14 | 19
  CXCL10 at baseline | 14195.394 (37588.5073) | 28501.304 (54928.0152) | 3654.197 (7505.8959)
  CXCL10 at EOT/Week 8: number analyzed (Participants) | 31 | 13 | 18
  CXCL10 at EOT/Week 8 | 3203.194 (13239.6238) | 6355.428 (20287.7247) | 926.580 (2389.4231)
  CXCL9 at baseline: number analyzed (Participants) | 34 | 15 | 19
  CXCL9 at baseline | 14113.999 (34451.6041) | 26695.379 (49400.5090) | 4181.331 (6470.0963)
  CXCL9 at EOT/Week 8: number analyzed (Participants) | 31 | 13 | 18
  CXCL9 at EOT/Week 8 | 2109.078 (10100.8802) | 4749.055 (15555.8338) | 202.428 (240.9550)
  sCD25 at baseline: number analyzed (Participants) | 34 | 15 | 19
  sCD25 at baseline | 17026.171 (13537.8951) | 23980.603 (13267.5834) | 11535.830 (11268.1072)
  sCD25 at EOT/Week 8: number analyzed (Participants) | 31 | 13 | 18
  sCD25 at EOT/Week 8 | 9882.585 (8542.0418) | 11301.162 (8847.8000) | 8858.058 (8417.5485)

18. Other Pre Specified Outcome: Number of Patients Who Demonstrated a Presence of Circulating Antibodies Against Emapalumab to Determine Immunogenicity
Description: The presence of circulating antibodies against emapalumab was inferred by positive results for anti-drug antibodies (ADAs).
Time Frame: Up to 1 year follow up post end of treatment with assessments at first dose of emapalumab, Week 4, Week 8, EOT and following treatment at day 100 and at the 1 year follow up visit, with data presented at study day 21 and EOT/Week 8.
Population: Number of patients who demonstrated a presence of circulating antibodies shown only for visits where a positive result was recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | All-treated Analysis Set | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced
Number analyzed (Participants) | 35 | 16 | 19
Participants
  Presence of circulating antibodies at Study Day 21 | 2 | 2 | 0
  Presence of circulating antibodies at End of Treatment/Week 8 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Signing of ICF until end of long-term follow-up (1 year after either HSCT or the last emapalumab infusion if HSCT was not performed). Through study completion. The average time 285 days.
Groups:
- All-treated Analysis Set - Treatment Experienced: Patients in the All-treated analysis set who could have received conventional HLH therapy without having obtained a satisfactory response according to the Investigator or having shown signs of intolerance to previous HLH therapy.
Arm/Group | All-treated Analysis Set - Treatment naïve | All-treated Analysis Set - Treatment Experienced | All-treated Analysis Set
All-Cause Mortality (participants affected / at risk) | 7/16 | 9/19 | 16/35
Serious Adverse Events (participants affected / at risk) | 16/16 | 16/19 | 32/35
Other Adverse Events (participants affected / at risk) | 14/16 | 19/19 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-treated Analysis Set - Treatment naïve (N=16) | All-treated Analysis Set - Treatment Experienced (N=19) | All-treated Analysis Set (N=35)
Condition aggravated (General disorders) | 4 (4) | 8 (8) | 12 (12)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 4 (4) | 5 (5)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 5 (5)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 2 (3) | 3 (4)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Herpes simplex viraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 4 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 3 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Engraftment syndrome (Immune system disorders) | 2 (2) | 1 (1) | 3 (3)
Acute graft versus host disease (Immune system disorders) | 2 (2) | 0 (0) | 2 (2)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Graft loss (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Fanconi syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Visual field defect (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-treated Analysis Set - Treatment naïve (N=16) | All-treated Analysis Set - Treatment Experienced (N=19) | All-treated Analysis Set (N=35)
Vomiting (Gastrointestinal disorders) | 7 (10) | 10 (15) | 17 (25)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 10 (16) | 15 (23)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 5 (6) | 7 (11)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 4 (7) | 6 (9)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 4 (5)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Anal erythema (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Anal blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 6 (11) | 8 (17) | 14 (28)
Pain (General disorders) | 3 (7) | 6 (9) | 9 (16)
Mucosal inflammation (General disorders) | 1 (1) | 4 (4) | 5 (5)
Oedema peripheral (General disorders) | 2 (2) | 2 (5) | 4 (6)
Condition aggravated (General disorders) | 2 (2) | 1 (1) | 3 (3)
Hypothermia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Catheter site rash (General disorders) | 0 (0) | 1 (1) | 1 (1)
Crying (General disorders) | 1 (2) | 0 (0) | 1 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vascular device occlusion (General disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (7) | 8 (13)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (7) | 4 (7)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 3 (4) | 1 (2) | 4 (6)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 3 (4) | 4 (5)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (3) | 3 (4)
Candida infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 3 (4)
Adenovirus reactivation (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Epstein-Barr virus infection reactivation (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Oral fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Paronychia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (4) | 1 (4)
Bacterial sepsis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis viral (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis neonatal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0) | 1 (3)
Adenovirus test positive (Investigations) | 1 (1) | 2 (3) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
C-reactive protein increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Weight increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Fibrin D dimer increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Gram stain positive (Investigations) | 0 (0) | 2 (2) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Human rhinovirus test positive (Investigations) | 0 (0) | 2 (2) | 2 (2)
Respirovirus test positive (Investigations) | 0 (0) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Candida test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Culture (Investigations) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Enterobacter test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Epstein-Barr virus test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glycocholic acid increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Pseudomonas test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Sapovirus test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Ultrasound abdomen abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Ultrasound kidney abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Ultrasound liver abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Vitamin D increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 5 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Interstitial lung abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6) | 7 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (4)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (4)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 5 (5) | 11 (11)
Hypotension (Vascular disorders) | 2 (2) | 1 (2) | 3 (4)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Venoocclusive disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 3 (4)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 4 (4) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 3 (5) | 4 (6)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Hypotonia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Cerebral ventricle dilatation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1) | 4 (4)
Nephrocalcinosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Kidney enlargement (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 1 (1) | 2 (2)
Acute graft versus host disease in intestine (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Cell-mediated immune deficiency (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Gallbladder oedema (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Anal injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 3 (4)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Genital injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 2 (2) | 4 (4)
Adrenal suppression (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Eyelid oedema (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Lagophthalmos (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Pain management (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Vitamin supplementation (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT03312751/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03312751/SAP_001.pdf